# Evaluation of treatment duration of En-masse versus Two steps Retraction in Patients having Maxillary Protrusion: A Randomized Clinical Trial

#### Consent form

Faculty of Oral and Dental Medicine, Future University in cairo

Submitted by

Aya Ahmed El Ashwal

B.D.S. Misr International University, 2012 (2019)



# RESEARCH ETHICS COMMITTEE Faculty of Oral and Dental Medicine (REC-FODM) CONSENT FORM (#3)

# Part I – Research Participant Information Sheet:

- A. Purpose of the Research: to determine which technique en-masse or two steps retraction shorter in treatment duration.
- B. Description of the Research: this trial will involve extraction of the first permanent premolars of the upper jaw in order to bring back the front teeth to correct procumbency of the lips and jaw.
- C. Potential Risks and Discomforts: pain associated with tooth movement, Undesired tooth movement, Root resorption
- D. Potential Benefits: orthodontic treatment is done for the patient as indicated, improving patients' esthetics, function and psychology including protrusion and procrumbency reduction.
- E. Cost: To participate in the research you will bear no additional costs or extra loss.

| | Document is approved for use by the cs Committee of FUE/FODM |
|---|---|
| Date From: _ | |
| To: | |



#### F. Compensation / Treatment:

In the event of injury resulting from participation in this research study, Researcher will make a treatment to you, its facilities and professional attention. Financial compensation from FUE/FODM is not available.

#### **G.** Voluntary Participation:

Participation in this study is voluntary. You will suffer no penalty nor loss of any benefits to which you are otherwise entitled should you decide not to participate. Withdrawal from this research study will not affect your ability to receive alternative methods of Dental care available at FUE/FODM. Significant new findings developed during the course of the research study which might be reasonably expected to affect your willingness to continue to participate in the research study will be provided

#### H. Confidentiality:

Your identity and medical record, as a participant in this research study, will remain confidential with respect to any publications that may result from this study. Furthermore, your Dental/medical record may be reviewed by the Research Advisory Council or the agency sponsoring this research in accordance with applicable laws and regulations.

| I. | Contact Person(s): |
|----|----------------------------------------------|
| | signed copy of the consent form will be give |

| | Document is approved for use by the ics Committee of FUE/FODM |
|---|---|
| Date From: | |
| To: | |



# PART II - Authorization for performance of certain procedures:

- 1. I/surrogate authorize Dr. Aya Ahmed El Ashwal and her associates to administer the following drugs, use the following devices or perform the following procedures during my treatment (or the treatment of the person named above for whom I am responsible)
- 2. I acknowledge that I have read, or had explained to me in a language I understand, the attached Research Participant Information sheet and that Dr Ava Ahmed El Ashwal has explained to me the nature of the procedures described in the Research Participant Information Sheet as well as any benefits to be expected, possible alternative methods of treatment, the attendant discomforts and risks reasonably to be expected and the possibility that complications from both known and unknown causes may arise as a result thereof. I was given ample opportunity to comprehensively inquire about this study and procedures and all my questions were answered to my satisfaction.
- 3. I understand that I am not entitled for reimbursement for expenses incurred as a result of my participation in this study

| | Document is approved for use by the ics Committee of FUE/FODM |
|------------|---------------------------------------------------------------|
| Date From: | |
| To: | |



- 4. I voluntarily accept the risks associated with the above-mentioned procedures with the knowledge and understanding that the extent to which they may be effective in my treatment (or the treatment of the patient named above, as the case may be) has not been established, that there may be side effects and complications from both known and unknown causes and that these procedures may not result in cure or improvement.
- 5. I understand that I am free to withdraw this consent and discontinue treatment with the above procedures at any time. The consequences and risks, if any, which might be involved in the event I later decide to discontinue such treatment, have been explained to me adequately. I understand that such withdrawal will not affect my ability to receive any dental/medical care made necessary by the performance of such studies or to which I might be otherwise entitled.
- the foregoing authorization and that all blanks or statements requiring completion were properly completed before I signed.

  Patient
  Name:
  File #:
  Patient/Surrogate:

  Signature

  Date

6. I confirm that I have read, or had read to me,

| This Consent Document is approved for use by the Research Ethics Committee of FUE/FODM REC #: | _ |
|---|---|
| Date From: | |
| To: | |

**Relationship:** 



7. I confirm that I have accurately translated and/or read the information to the subject or his/her surrogate.

| ms/ner surrogate. | | |
|---|---|---|
| Name: | | |
| Signature: | | |
| FUE ID #: Date: | - | |
| 8. I have fully explained to the above patient/ relative/ guardian the nature and purpose of the foregoing procedures, possible alternative methods of treatment which might be advantageous, the reasonable benefits to be expected, the attendant discomforts and risks involved, the possibility that complications may arise as a result thereof and the consequences and risks, if any, which might be involved in the event the patient/ relative/ guardian hereafter decides to discontinue such treatment. It is my understanding that the above patient/ relative/ guardian understand the nature, purposes, benefits, and risks of participation in this research before signing of this informed consent. I have also offered to answer any questions the above patient/ relative/ guardian might have with respect to such procedures and have fully and completely answered all such questions. | | |
| (Signature of Principal Investigator/ Delegate): | | <br>: |
| This Consent Document is approved for use by the Research Ethics Committee of FUE/FODM REC #: Date From: To: | | |



| UNIVERSITY IN EGYPT | |
|---|---|
| Research Ethics Committees Faculty of Oral and Dental Medicine | |
| Print Name: Aya Ahmed El Ashwa | l |
| Title: Master Student at FUE | |
| Date: | |
| This Consent Document is approved for use by the Research Ethics Committee of FUE/FODM | |
| REC # : | - |
| To: | |